CLINICAL TRIAL: NCT04334655
Title: Effects of Physical Therapy on Isometric Neck Retraction Strength and Pain in Patients With Neck Disability
Status: Completed | Type: Observational
Sponsor: Campbell University, Incorporated (Other)
Responsible Party: Principal Investigator, Frank Tudini, Assistant Professor, Campbell University, Incorporated
Other Study IDs: CampbellU
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Neck Pain; Strength
Keywords: Neck Pain; Strength; Physical Therapy
MeSH Terms: conditions — Neck Pain | interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Clinic 1: Clinics will be identified using Clinic numbers: Clinic 1, Clinic 2, Clinic 3, Clinic 4. The interventions will be normal physical therapy interventions. The only addition is the monitoring of isometric neck retraction strength at the initial evaluation, progress reports, and discharge. The purpose of the study is not to administer new or specific interventions but to monitor neck strength changes over time during regular physical therapy care.
  Interventions: Other: Physical Therapy
- Clinic 2: Clinics will be identified using Clinic numbers: Clinic 1, Clinic 2, Clinic 3, Clinic 4. The interventions will be normal physical therapy interventions. The only addition is the monitoring of isometric neck retraction strength at the initial evaluation, progress reports, and discharge. The purpose of the study is not to administer new or specific interventions but to monitor neck strength changes over time during regular physical therapy care.
  Interventions: Other: Physical Therapy
- Clinic 3: Clinics will be identified using Clinic numbers: Clinic 1, Clinic 2, Clinic 3, Clinic 4. The interventions will be normal physical therapy interventions. The only addition is the monitoring of isometric neck retraction strength at the initial evaluation, progress reports, and discharge. The purpose of the study is not to administer new or specific interventions but to monitor neck strength changes over time during regular physical therapy care.
  Interventions: Other: Physical Therapy
- Clinic 4: Clinics will be identified using Clinic numbers: Clinic 1, Clinic 2, Clinic 3, Clinic 4. The interventions will be normal physical therapy interventions. The only addition is the monitoring of isometric neck retraction strength at the initial evaluation, progress reports, and discharge. The purpose of the study is not to administer new or specific interventions but to monitor neck strength changes over time during regular physical therapy care.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Patients with primary complaints of neck pain will receive routine physical therapy care including modalities, manual therapy including neck mobilization and manipulation, stretching and strengthening exercises, and patient education.
  Other Names: Rehabilitation; Neck Strengthening

SUMMARY:
Impaired neck muscle strength is related to neck pain, abnormal posture, and various cervical pathologies. Clinicians, therefore require objective, reliable and valid methods for quantifying neck strength. In a previous study, the investigators developed a novel, valid, and reliable method for measuring neck retraction strength, using a handheld dynamometer (HHD), in normal, healthy individuals. The investigators are now expanding this research to study a patient population. Specifically, to describe isometric neck retraction strength in patients with neck pain and to study the effects of physical therapy (PT) on that strength. Our hypothesis is that isometric cervical retraction strength will increase over the course of treatment and that there will be an inverse relationship between strength and the Numeric Pain Rating Scale (NPRS) and Neck Disability Index (NDI).

DETAILED DESCRIPTION:
Four physical therapists from four different outpatient clinics will collect demographic, anthropomorphic, and isometric neck retraction strength data with an HHD in patients with primary complaints of neck pain at the time of the initial evaluation, regular follow-ups, and at discharge. The PT will also include a shortlist of the primary interventions used during the course of treatment. A short video explaining how to test isometric neck retraction strength will be provided to each clinic and the description can also be found in the investigator's previous article entitled "Reliability and validity of measurements of cervical retraction strength obtained with a hand-held dynamometer." Basically, the patient will lay on their back with the HHD under the external occipital protuberance. The patient will then perform a practice isometric contraction at 50% maximum force followed by two maximum effort trials with 1-minute in-between.

A follow-up phone call will be made to each clinic to assure that the units arrived and to answer any additional questions regarding the procedure or data to be collected. Follow up phone calls will then be performed monthly to assess progress. At the end of three months, a preliminary analysis, based on the total number of documented patients will be made. A power analysis indicates that 40 patients will be sufficient to answer our research question. This is based on a 2007 article by Cagnie, B. in the Archives of Physical Medicine Rehabilitation entitled "Differences in isometric neck muscle strength between healthy controls and women with chronic neck pain: the use of a reliable measurement." To account for drop-outs the investigators raised this to an n=60.

Data will be collected over a secure Qualtrics server to which each participating PT will have an individual access code. No identifiable patient information will be given to the investigators. Data analysis will include Pearson or Spearman correlation coefficients to examine the relationship between isometric neck strength with patient-reported outcome measures including the Numeric Pain Rating Scale (NPRS) and Neck Disability Index (NDI). Repeat Measure ANOVA will be used to compare the variables including strength over different time frames throughout the episode of care. An intention to treat analysis will be used for patients who do not complete the study or their Physical Therapy (PT) care.

Data will be collected on 60 consecutive patients with neck pain. Inclusion criteria include patients over the age of 18 years that are receiving physical therapy with primary complaints of neck pain. Exclusion criteria include individuals with a history of cervical neck surgery as well as those with neurologic diseases or Chronic Obstructive Pulmonary Disease (COPD).

Day 1: Patient with a primary complaint of neck pain is seen in one of the four physical therapy clinics participating in the study. The patient is recruited by the PT in the clinic. The study will be explained to the patient and written consent obtained and filed in the clinic. A copy of the consent will also be given to the participant.

The PT conducts their initial evaluation and treatment as they normally would with the addition of a test for isometric neck strength. Measuring neck strength is a normal procedure for a PT to perform and is well within the scope of practice for physical therapists. Many clinics do not have hand-held dynamometers (HHD) so we will be providing the dynamometers and mailing them to each clinic. The MicroFET2 hand-held dynamometer is FDA approved (Regulation number: 21 CFR 888.1240) and will be used only in the manner for which it was attended, i.e. to measure isometric strength. The hand-held dynamometer is placed in a cradle behind the patient's head in supine. Instructions are given to retract the chin and head into the dynamometer three times. 1 practice trial at 50% and 2 maximum effort trials with 1 minute between attempts. This is outlined in the investigator's 2019 study (Reliability and validity of measurements of cervical retraction strength obtained with a hand-held dynamometer. Journal of Manual and Manipulative Therapy. 2019;27(4): 222-228.) The entire procedure will take approximately 5 minutes. This information is recorded along with anthropomorphic data, pain levels, neck disability index, and treatment performed. All information is coded and sent to the primary researchers over a secure Qualtrics connection.

4. The patient will receive regular Physical Therapy care. The neck strength, pain, and neck disability index are recorded at re-assessments (usually monthly) and at discharge. The use of this assessment will in no way impact the quality or quantity of PT received by the patient.

ELIGIBILITY:
Inclusion Criteria:

- 18 years of age or older Primary complaints of neck pain and receiving Physical Therapy

Exclusion Criteria:

- History of neck surgery Neurologic diseases Chronic Obstructive Pulmonary Disease (COPD)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with neck pain receiving physical therapy
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2021-10-23 (Actual)

PRIMARY OUTCOMES:
Change in Neck Retraction Strength | At baseline (the initial evaluation) and every 30 days thereafter until discharge from PT. The estimated period of time from baseline until completion is 3 months.
  Change in isometric Neck Retraction Strength measured with a Hoggan MicroFET2 hand-held dynamometer in kilograms at baseline, approximately every 30 days during the physical therapy intervention and immediately after the physical therapy intervention at discharge. The estimated period of time from baseline until completion is 3 months.

SECONDARY OUTCOMES:
Change in Neck Pain: Numeric Pain Rating Scale (NPRS) | At baseline (the initial evaluation) and every 30 days thereafter until discharge from PT. The estimated time frame from baseline until completion is 3 months.
  Change in subjective reports of neck pain on the Numeric Pain Rating Scale (NPRS) will be recorded by the physical therapist for each subject on a 0 - 10 point scale with "0" being no pain and "10" being extreme pain or the worst pain imaginable. The pain level will be recorded at baseline, approximately every 30 days during the physical therapy intervention, and immediately after the physical therapy intervention at discharge. The estimated time frame from baseline until completion is 3 months.
Function | At baseline (the initial evaluation) and every 30 days thereafter until discharge from PT. The estimated time frame from baseline until completion is 3 months.
  Change in Neck Disability Index (NDI) Score. The Neck Disability Index is a patient reported outcome measure that will be completed by each participant at baseline, approximately every 30 days during the physical therapy intervention and immediately after the physical therapy intervention at discharge. The questionnaire is reported as a percentage (%) with higher scores indicating higher levels of disability. The estimated time frame from baseline until completion is 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Tudini, DSc, Principal Investigator — Campbell University
Locations (4):
- United States (4):
  - Integral Physical Therapy, Firestone, Colorado
  - Performance PT, Cos Cob, Connecticut
  - Connecticut Physical Therapy Specialists, Granby, Connecticut
  - Back in Action, Holly Springs, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
Data will be de-identified in each clinic and then shared with the primary investigator at Campbell University. The de-identified data will be available after data analysis is performed.

REFERENCES:
- [Result] Tudini F, Myers B, Bohannon R. Reliability and validity of measurements of cervical retraction strength obtained with a hand-held dynamometer. J Man Manip Ther. 2019 Sep;27(4):222-228. doi: 10.1080/10669817.2019.1586167. Epub 2019 Mar 18. PMID 30935321
- [Result] Cagnie B, Cools A, De Loose V, Cambier D, Danneels L. Differences in isometric neck muscle strength between healthy controls and women with chronic neck pain: the use of a reliable measurement. Arch Phys Med Rehabil. 2007 Nov;88(11):1441-5. doi: 10.1016/j.apmr.2007.06.776. PMID 17964885

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT04334655/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT04334655/ICF_002.pdf